CLINICAL TRIAL: NCT07065227
Title: Potential Benefits of Sonic Augmentation Technology in Music for Improving Health and Wellness
Brief Title: Potential Benefits of Sonic Augmentation Technology in Music
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Keeping the study open for future recruitment.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB202500959
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-07

CONDITIONS: Biobehavioral State; Sonic Augmentation Technology; Oxytocin; Autonomic Reactivity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the augmented or control music group. Both groups will complete a pre-survey and provide a saliva sample. Following the 15-minutes of music, participants will provide a saliva sample and complete a post-survey.
Who Masked: Participant
Masking Description: Participants will be randomly assigned via a random number generator to either the augmented group or the control group. The participant will be blinded to the group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Theme (Experimental): Participants complete the pre-survey, and provide 1.5-2mL of saliva. After that, the participants will receive 15-minutes of the augmented music. After completion of the music, Study Staff will have the participants provide 1.5-2mL of saliva and complete the post-survey.
  Interventions: Behavioral: Augmented Theme
- Mozart Theme (Active Comparator): Participants complete the pre-survey, and provide 1.5-2mL of saliva. After that, the participants will receive 15-minutes of the control music featuring a Mozart composition. After completion of the music, Study Staff will have the participants provide 1.5-2mL of saliva and complete the post-survey.
  Interventions: Behavioral: Mozart Theme

INTERVENTIONS:
Behavioral: Augmented Theme — The music is augmented by embedding the natural rhythms of bodily functions (e.g. breathing, heart rate variability, vascular tone, etc) that signal the body to calm.
  Arms: Augmented Theme
Behavioral: Mozart Theme — The selected Mozart composition consists of: Composition Eine kleine Nachtmusik, K. 525 (5 minutes 30 seconds), Andante from Piano Concerto No. 21, K. 467 (6 minutes 30 seconds), and Ave verum corpus, K. 618 (3 minutes).
  Arms: Mozart Theme

SUMMARY:
The goal of this clinical trial is to explore possible benefits and mechanisms through which listening to music enhanced with Sonic Augmentation Technology (SAT) can improve health and wellness. The main goals of the study are:

* To examine the immediate effects of listening to the augmented music.
* To identify individual characteristics that influence the immediate effects of listening to the augmented music.

Participants will:

* Complete the online pre- and post-surveys.
* Provide pre- and post- music saliva samples (1.5mL).
* Listen to the full 15-minutes music session via over-ear headphones.

DETAILED DESCRIPTION:
The purpose of the current study is to explore the effects of listening to 15-minutes of sonic augmented music on subjective feelings of calmness and autonomic state.

Specific Aims:

Specific Aim 1: To investigate whether pre-intervention measures of current functioning relate to the overall functioning of the participants.

•The investigators will examine measures of autonomic reactivity to prior mental health and medical adversity, embodiment, and emotional and physical health.

Specific Aim 2: To identify the immediate effects of listening to the music

•The investigators will explore whether listening to the music leads to improvements in the functioning. First, the investigators will compare the participants who listened to the SAT enhanced music to the participants who listened to the Mozart composition (control).

Specific Aim 3: To identify individual characteristics that influence the effectiveness of listening to the SAT music immediately •The investigators will explore the impact of specific vulnerability and resiliency factors (e.g., prior mental and medical adversity) on how well participants benefit from listening to the music immediately.

Specific Aim 4: To investigate levels of oxytocin after listening to the music.

•The investigators will explore whether listening to SAT enhanced music leads to changes in oxytocin. Specifically, we will compare the levels of salivary oxytocin before and after the intervention in two groups: participants who listen to 15 minutes of the Mozart theme and participants who listen to 15 minutes of the augmented theme.

Experimental design

* The participants will be randomly assigned to either the augmented music group or the control group featuring a Mozart composition.

  * Augmented music group: The music is augmented by embedding the natural rhythms of bodily functions (e.g. breathing, heart rate variability, vascular tone, etc) that signal the body to calm.
  * Control group: The selected Mozart composition consists of: Composition Eine kleine Nachtmusik, K. 525 (5 minutes 30 seconds), Andante from Piano Concerto No. 21, K. 467 (6 minutes 30 seconds), and Ave verum corpus, K. 618 (3 minutes). This composition is structured to serve as emotionally immersive, musically coherent control conditions in a 15-minute experimental paradigm.
* The control group will listen to 15 minutes of control music, and the augmented group will listen to 15 minutes of augmented music.
* At pre- and post-, the participants will complete online self-report surveys and provide 1.5mL of saliva.
* Between-subject analyses will compare those who listened only to the augmented 15-minute music sample and those who listened to the control 15-minutes of music to determine if those who listened to the augmented music exhibit greater changes than those who did not. Subject analyses will determine the potential benefits of listening to music for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 89
* Proficient in English
* Employed at UF Health Jacksonville

Exclusion Criteria:

•Over the age of 89

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Assessing the Impact of Autonomic Reactivity using the Body Perceptions Inventory Short Form | Baseline
  This 20-item measure is scored on a 5-point Likert scale (never = 1, occasionally = 2, sometimes = 3, usually = 4, always = 5). Items are summed to determine total autonomic reactivity score, with the higher scores indicating greater autonomic reactivity
Assessing the Impact of Adversity History on the Effectiveness of Listening to Music | Baseline
  This measure assesses the impact of six types of traumatic experiences (childhood adverse experiences, childhood maltreatment, intimate partner maltreatment, other person maltreatment, life-threatening situations, sudden losses, and person health situations). Each item is scored on a 5-point Likert scale (did not occur = 0, occurred and no impact on my life = 1 to big impact on my life = 4). Items are summed to determine total impact scores.
Measuring Change in subjective feelings of calmness and autonomic state using the Benefits List | From baseline through study completion, an average of 90 minutes
  This 12-item measure, which assesses subjective feelings of calmness and autonomic state was created for this study.
Assessing the Impact of anxiety on the Effectiveness of Listening to Music using the GAD-7 | Baseline
  This 7-item measure assesses the severity of generalized anxiety symptoms. It is scored on a 4-point Likert scale (not at all = 0, several days = 1, more than half the days = 2, nearly every day = 3). The items are summed to calculate the total anxiety score, with higher scores indicating more severe anxiety symptoms.
Assessing the Impact of depression on the Effectiveness of Listening to Music using the PHQ-8 | Baseline
  This 8-item measure assesses the severity of depressive symptoms. It is scored on a 4-point Likert scale (not at all = 0, several days = 1, more than half the days = 2, nearly every day = 3). The items are summed to determine the total depression score, with higher scores indicating greater severity of depressive symptoms.
Assessing the Impact of PTSD on the Effectiveness of Listening to Music using the PCL-5 | Baseline
  This 8-item measure assesses the severity of depressive symptoms. It is scored on a 5-point Likert scale (not at all = 0, a little bit = 1, moderately = 2, quite a bit = 3, 4 = extremely). The items are summed to determine the total PTSD score, with higher scores indicating greater severity of PTSD symptoms.
Assessing the Impact of Moral Injury on the Effectiveness of Listening to Music using the Moral Injury Events Scale | Baseline
  This 6-item measure assesses the level of agreement about the occurrence and anguish of moral injury (asked as two separate questions) experienced by participants themselves (self moral injury or Self MI) and observed by participants in others (others moral injury or Others MI). It is scored on a 5-point Likert scale (strongly disagree = 1, Moderately Disagree = 2, 3 = disagree, 4 = agree, 5 = moderately agree, 6 = strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes P. Dale, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville Wellness Center Building, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to protect the privacy of participants.